CLINICAL TRIAL: NCT04737278
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Study Evaluating the Safety and Efficacy of Cunermuspir on Energy, Strength, Fatigue and Discomfort in Subjects With Nerve or Muscle Pain
Brief Title: Safety and Efficacy of Cunermuspir on Energy, Strength, and Fatigue in Patients With Nerve or Muscle Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mitosynergy LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13MFHM
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Neuralgia; Myalgia
Keywords: Copper; nicotinic acid; energy; strength; fatigue; nerve pain; muscle pain; neuralgia; myalgia
MeSH Terms: conditions — Neuralgia; Myalgia; Fatigue

STUDY DESIGN:
Intervention Model Description: randomized, double--blind, placebo controlled, parallel study
Who Masked: Participant, Investigator
Masking Description: The investigational product bottles were labeled according to the requirements of ICH--GCP guidelines and applicable local regulatory guidelines. Investigational products were coded by the unblinded personnel at KGK Synergize who were not involved in the collecting or analyzing of study data. Each package contained a similar label differing only in randomization number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cunermuspir (Experimental): Cunermuspir (Copper Niacin Chelate) 6.06mg per capsule. Non--medicinal ingredients: Organic evaporated cane juice powder, hypromellose, titanium dioxide Two doses per day: one with the morning meal and the other with a mid afternoon snack. The study duration was 28 days.
  Interventions: Drug: Cunermuspir
- Placebo (Placebo Comparator): Organic evaporated cane juice powder, hypromellose, titanium dioxide. Same dosing as Cunermuspir arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cunermuspir — Copper Niacin Chelate, 6.06 mg per capsule Non-medicinal ingredients:
  Organic evaporated cane juice powder, hypromellose, titanium dioxide
  Other Names: cuprous nicotinic acid
  Arms: Cunermuspir
Other: Placebo — same non-medical ingredients and encapsulation as Intervention 1
  Arms: Placebo

SUMMARY:
Male and female participants were selected based on chronic neuromuscular pain. Patients were instructed to take two doses of the placebo or cuprous nicotinic acid chelate Cunermusmir twice a day for 28 days. Hypothesis: Cunermuspir would improve quality of life as determined by several questionnaires.

DETAILED DESCRIPTION:
A total of 72 subjects were consented and screened, with 56 subjects (28 males and 28 female) being eligible to participate in the study. Fifty-six subjects with muscle/nerve pain were randomized at a ratio of 1:1 to one of two treatment groups. To evaluate primary and secondary objectives, study assessments were conducted at Baseline, and Day 28 ± 2. The Individualized Neuromuscular Quality of Life Questionnaire (INQoL), Symptom Impact Questionnaire (SQIR), Mini-Mental State Examination (MMSE) were completed by participants to assess physical function, pain, fatigue/energy and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-75
* If female, subject is not of child bearing potential. Defined as females who have
* had a hysterectomy or oophorectomy.
* bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).
* Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include: Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo--Provera, Lunelle), or hormone implant (Norplant System), Intrauterine devices, Vasectomy of partner, Total Abstinence
* Subject has unresolved persistent muscle or nerve pain (muscle or nerve pain population)
* Subjects using other therapies for nerve/muscle pain (e.g., exercise, TENS, acupuncture, exercise, psychotherapy, massage, physiotherapy, etc), must be used at a stable schedule for 1 month prior to the trial and subject agrees to continue these therapies at the same schedule during the trial avoiding changes in frequency or intensity and to record therapies in the study diary
* Agrees to comply with study procedures
* Has given voluntary, written, informed consent to participate in
* the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Planned surgery during the course of the trial
* Use of prescription drugs for fibromyalgia or nerve pain (e.g.Lyrica, Cymbalta and Savella and others).
* Use of prescription medications for depression, anxiety or other mental disorders
* Requires the use of prescription drugs to control pain (other than provided rescue medication)
* Use of oral or topical prescription or over the counter medications or natural health products for pain relief 3 days prior to randomization and during the trial (other than provided rescue medication)
* Use of natural health products including vitamins and minerals within 3 days prior to randomization and during the trial
* Use of blood thinning medications (e.g. warfarin)
* Chronic lyme disease or chronic parasitic infections
* Uncontrolled hypertension defined as untreated systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg
* Subjects with diabetes
* History of bleeding disorders, or significant blood loss in the past 3 months
* Alcohol use >2 standard alcoholic drinks per day and/or alcohol or drug abuse within the past year
* Allergy or sensitivity to study supplement ingredients or acetaminophen
* Participation in a clinical research trial within 30 days prior to randomization
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2014-05-28 (Actual); Study Completion 2014-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Synergize now KGK Science, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Close collaboration with KGK Synergize/Science will be needed to determine which data can be legally shared. In retrospective analysis of data six years later, raw data in the form of a spreadsheet proved to be extremely valuable.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be shared as soon as Mitosynergy meets the regulatory requirements for sharing.
Access Criteria: Access will be determined by regulatory requirements. Mitosynergy favors as broad access as the law allows. If the law permits access on company websites, Mitosynergy will favor this.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 met the enrollment requirements. Of these only 49 completed the study
Groups:
- Cunermuspir: Cunermuspir (Copper Niacin Chelate) 6.06mg per capsule. Non--medicinal ingredients: Organic evaporated cane juice powder, hypromellose, titanium dioxide Two doses per day: one with the morning meal and the other with a mid afternoon snack. The study duration was 28 days.
  Cunermuspir: Copper Niacin Chelate, 6.06 mg per capsule Non-medicinal ingredients:
  Organic evaporated cane juice powder, hypromellose, titanium dioxide
Period: Overall Study
Arm/Group | Cunermuspir | Placebo
Started | 28 | 28
Completed | 24 | 25
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — failure to complete questionnaire | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cunermuspir | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.6) | 48.2 (10.4) | 46.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  Canada | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Neuromuscular Symptoms
Description: Quality of life was assessed by using the Individualized Neuromuscular Quality of Life Questionnaire (INQoL) Answers to symptom questions are scored from 0 to 6 or 7 with 0 being "none at all" and and 6 to 7 being "an extreme amount" There are three questions regarding pain. The pain score is (a+b+c)/19 x100. The higher the score, the greater the symptom impact.
Time Frame: baseline and 28 days after enrollment
Population: Three patients were lost to followup.Four other patients had testing issues that the study investigators deemed them to be removed from baseline and day 28 analyses. This is why there are not 28 patients represented in baseline whereas there are in toxicology related outcome measures.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 24 | 25
score on a scale
  baseline | 36.5 (16.4) | 43.5 (21.1)
  Day 28 | 28.5 (18.6) | 32.7 (23.0)
Statistical Analysis 1: Comparison: Placebo; Test type: Other — test of the hypothesis that the score on day 28 is different from the baseline score in the Placebo group; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Cunermuspir; test of the hypothesis that the score on day 28 is different than the baseline score; Test type: Other; p = 0.01, t-test, 2 sided

2. Primary Outcome: Platelet ATP
Description: Platelet ATP levels were measured as previously published in the literature.
Time Frame: baseline and 28 days after enrollment
Population: ATP isolated from platelets. Some samples were not used for analysis due to contamination with red blood cells.
Measure: Mean (Standard Deviation); unit: nmol / E9 Platelets
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 21 | 25
nmol / E9 Platelets
  baseline | 43.6 (16.4) | 42 (13.1)
  day 28 | 59.2 (20.1) | 51.2 (15.0)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Day 28. Between group comparison was made using ANCOVA accounting for baseline values, no significance at p<0.05. Within group comparisons were made using the paired Student's t test; Test type: Other; p = 0.15, t-test, 2 sided

3. Secondary Outcome: Household Chores and Neuro Muscular Sumptoms
Description: Physical function in performing household chores was assessed using the Revised Symptom Impact Questionnaire (SQIR) For each household chore participants are asked to check 1 of 11 boxes between "no difficulty" and "extremely difficult" No difficulty is scored as 0 and extreme difficulty with the task is scored as 10. The higher the score, the more difficulty experienced performing the chore. Friend & Bennett Arthritis Res & Therapy 2011. Household chores are just one module with 9 questions for a maximum of 90 points. These scores are summed and divided by 3. Module 2 relates to the emotional impact with only two questions for a total of 20 points. Module 3 relates to physical symptoms with a total of ten questions worth a maximum of 100 points. This score is divided by 2. The three modules are summed for a total impact score of 100 points. A score of 0 indicates absolutely no impact and a score of 100 the greatest possible impact.
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 24 | 25
units on a scale
  baseline | 27.6 (16.8) | 34.9 (16.9)
  day 28 | 16.7 (10.9) | 29.3 (28.7)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p < 0.01, ANCOVA
Statistical Analysis 2: Comparison: Cunermuspir vs Placebo; comparison made between placebo and Cunermuspir at baseline; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cunermuspir vs Placebo; comparison made at day 28; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cunermuspir; comparison between baseline and day 28; Test type: Other; p = 0.07, t-test, 2 sided

4. Secondary Outcome: Cognition
Description: Cognition is the mental process of knowing, including aspects such as awareness, perception, reasoning, and judgment. The mini-mental state exam (MMSE) puts a number to "cognition." Any score of 24 or more out of a total 30 points is considered normal cognition. A test taker may be asked to orientate in space and time by recalling aspects of the physical location as well as month, day, year, and perhaps season. Simple mathematical calculations like counting backwards from 100 by seven may also be included. A complex command such as redrawing geometric figures scores six points in this exam. Since none of the participates were cognitively impaired, the investigators decided to make obtaining a perfect score on this exam an outcome measure.
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 1
Measure: Number; unit: participants with perfect score
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 24 | 25
participants with perfect score
  baseline | 18 | 16
  day 28 | 22 | 18
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; base line between group comparisons; Test type: Other; p = 0.54, Fisher Exact
Statistical Analysis 2: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.14, Fisher Exact

5. Secondary Outcome: Heart Rate
Description: heart rate is measured in beats per minute
Time Frame: baseline and 28 days after enrollment
Population: For toxicology outcome measures the investigators included all 28 participants in each group at baseline as well as data for the 26 (Cunermuspir) and 27 (Placebo) remaining at day 28. The investigators considered these data valid in spite of issues with the questionnaires of other outcome measures
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
beats per minute
  baseline | 70.3 (10.8) | 68.2 (8.1)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 68.3 (9.7) | 69.7 (9.4)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.54, ANCOVA

6. Secondary Outcome: Diastolic Blood Pressure
Description: The diastolic blood pressure was measured in mm Hg
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mm Hg
  baseline | 70.5 (6.4) | 75.0 (9.4)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 69.3 (7.3) | 74.6 (7.3)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; The original report from KGK Synergize/Science did not specify if the results are ANCOVA or a between group comparison at 2ay 28; Test type: Other; p < 0.01, ANCOVA

7. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure was measured in mm Hg
Time Frame: baseline and 28 days after enrollment.
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mm Hg
  baseline | 111.7 (10.6) | 114.6 (13.1)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 109.5 (15.8) | 112.3 (11.2)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.31, ANCOVA

8. Secondary Outcome: Hemoglobin
Description: changes measured in g/L blood
Time Frame: baseline and 28 days after enrollment.
Population: as for outcome 5
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
g/L
  baseline | 140.3 (12.9) | 141.3 (12.4)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 142.2 (14.3) | 141.0 (12.0)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.48, ANCOVA

9. Secondary Outcome: Hematocrit
Description: changes in the fraction of whole blood occupied by red blood cells measured as L/L
Time Frame: baseline and 28 days after enrollment
Population: Three participants were lost to followup on day 28. For toxicology outcome measures the investigators included all 28 participants in each group at baseline as well as data for the 26 (Cunermuspir) and 27 (Placebo) remaining at day 28. The investigators considered these data valid in spite of issues with the questionnaires of other outcome measures
Measure: Mean (Standard Error); unit: L/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
L/L
  baseline | 0.411 (0.034) | 0.416 (0.032)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 0.416 (0.038) | 0.415 (0.031)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.84, ANCOVA

10. Secondary Outcome: WBC
Description: changes in white blood cells (WBC) measured in units of 10^9 per liter blood
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^9 cells/L
  baseline | 5.93 (1.57) | 5.82 (1.50)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 5.88 (1.81) | 6.00 (1.34)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.63, ANCOVA

11. Secondary Outcome: RBC
Description: changes in red blood cells (RBC) measured in units of 10^12 per liter blood
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: 10^12 cells/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^12 cells/L
  baseline | 4.76 (0.38) | 4.74 (0.38)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 4.82 (0.41) | 4.73 (0.38)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.05, ANCOVA

12. Secondary Outcome: MCV
Description: changes in mean corpuscular volume (MCV) measured in units of fL
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fempto liter per cell
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
fempto liter per cell
  baseline | 86.2 (3.9) | 87.7 (3.1)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 86.4 (4.3) | 87.7 (3.1)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p < 0.01, ANCOVA

13. Secondary Outcome: MCH
Description: changes in mean corpuscular hemoglobin, measured in units of pg, the average amount of hemoglobin in a single RBC
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: pg per cell
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
pg per cell
  baseline | 29.5 (1.64) | 29.81 (1.36)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 29.48 (1.69) | 29.86 (1.29)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p < 0.01, ANCOVA

14. Secondary Outcome: MCHC
Description: mean corpuscular hemoglobin concentration is the concentration of hemoglobin in a single RBC measured in units of g/L
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
g/L
  baseline | 342.4 (8.2) | 339.9 (7.8)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 341.2 (6.4) | 340.5 (5.7)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.48, ANCOVA

15. Secondary Outcome: RDW
Description: changes in the RBC distribution width (RDW) are reported in units of percentage (%)
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: red cell distribution width %
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
red cell distribution width %
  baseline | 13.78 (0.70) | 13.80 (0.50)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 13.77 (0.63) | 13.93 (0.58)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.06, ANCOVA

16. Secondary Outcome: Platelets
Description: changes in the platelet counts are reported in units of 10^9 per liter blood
Time Frame: baseline and 28 days after enrollment
Population: By day 28 three participants were lost to followup: two in the Cunermuspir group and one in the placebo group. There were issues in handling of one platelet sample in the Cunermuspir group. This brings the number in the Cunermuspir group down to 25 on day 28. For technical reasons, platelet data are missing for subject 021. All other blood cell data are present in this report of data.
Measure: Mean (Standard Error); unit: 10^9 platelets/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^9 platelets/L
  baseline | 250 (62) | 266 (71)
  day 28: number analyzed (Participants) | 25 | 27
  day 28 | 255 (65) | 269 (69)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.02, ANCOVA

17. Secondary Outcome: Neutrophils
Description: changes in neutrophils are reported in units of 10^9 per liter blood
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^9 cells/L
  baseline | 3.28 (1.06) | 3.35 (1.13)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 3.15 (1.19) | 3.60 (1.13)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.03, ANCOVA
Statistical Analysis 2: Comparison: Placebo; comparison of neutrophils from baseline to day 28; Test type: Other; p = 0.05, t-test, 2 sided

18. Secondary Outcome: Lymphocyte
Description: changes in lymphocytes are reported in units of 10^9 per liter blood
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^9 cells/L
  baseline | 2.01 (0.64) | 1.83 (0.51)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 2.04 (0.72) | 1.74 (0.51)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p < 0.01, ANCOVA

19. Secondary Outcome: Monocyte
Description: changes in monocytes are reported in units of 10^9 per liter blood
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^9 cells/L
  baseline | 0.450 (0.137) | 0.475 (0.140)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 0.473 (0.176) | 0.500 (0.124)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; comparison of baseline values; Test type: Other; p = 0.47, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cunermuspir vs Placebo; comparison performed on data from day 28; Test type: Other; p = 0.24, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Eosinophil
Description: changes in eosinophils are reported in units of 10^9 cells per liter blood
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^9 cells/L
  baseline | 0.154 (0.074) | 0.143 (0.063)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 0.181 (0.110) | 0.130 (0.072)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; comparison of eosinophil counts at day 28; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Basophil
Description: changes in basophils are reported in units of 10^9 cells per liter blood
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
10^9 cells/L
  baseline | 0.0107 (0.0315) | 0.0071 (0.0262)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 0.0077 (0.0272) | 0.0074 (0.0267)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; The day 28 basophil counts on day 28 were compared between the two arms of this study; Test type: Other; p = 0.98, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: NLR
Description: Changes in the neutrophil to lymphocyte ratio (NLR) are reported as a dimensionless fraction of 1
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: dimensionaless units
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
dimensionaless units
  baseline | 1.77 (0.15) | 1.90 (0.13)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 1.67 (0.14) | 2.24 (0.19)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; All other statistical analyses were performed by KGK Synergize. This site was used to determine that the NLR were normally distributed https://www.gigacalculator.com/calculators/normality-test-calculator.php Because these data fulfilled the assumptions of ANOVA, the data were analyzed using this site: http://vassarstats.net/anova2u.html; Test type: Other; p = 0.025, ANOVA — This p value is for the treatment source. Visits (p=0.422) and visits x treatments (p=0.153) did not meet the threshold of significance

23. Secondary Outcome: Glucose
Description: changes in blood glucose are reported in units of mmol per liter
Time Frame: baseline and 28 days after enrollment
Population: In this population the initial screening was considered the baseline for all blood chemistry parameters. Three of the the participants were lost to followup or withdrew from the study
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mmol/L
  baseline | 5.12 (0.55) | 5.30 (0.42)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 5.25 (0.44) | 5.24 (0.48)
Statistical Analysis 1: Comparison: Cunermuspir; Comparison of blood glucose in the Cunermuspir arm between enrollment baseline and day 28; Test type: Other; p = 0.06, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; Comparison of enrollment baseline blood glucose and day 28 in the placebo arm; Test type: Other; p = 0.04, t-test, 2 sided
Statistical Analysis 3: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.92, ANCOVA

24. Secondary Outcome: Urea
Description: changes in renal function as measured by blood urea are reported in units of mmol per liter
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mmol/L
  baseline | 5.16 (1.13) | 5.33 (1.25)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 5.05 (1.57) | 5.26 (1.08)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.51, ANCOVA

25. Secondary Outcome: Creatinine
Description: changes in creatinine are reported in units of micromol per liter
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: micromol/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
micromol/L
  baseline | 72.2 (11.6) | 72.9 (16.0)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 72.3 (13.7) | 73.7 (15.0)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.38, ANCOVA

26. Secondary Outcome: eGFR
Description: changes in the estimated glomerular filtration rate (eGFR) are reported in units of mL/min/1.73m^2
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mL/min/1.73 m^2
  baseline | 90.4 (17.3) | 88.8 (16.2)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 91.2 (18.3) | 85.9 (15.7)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.01, ANCOVA

27. Secondary Outcome: Sodium
Description: changes in plasma sodium are reported in units of mmol per liter, reference range is 133-146 mEq/L, same as mM/L bloodbook.com
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mmol/L
  baseline | 143.39 (2.25) | 143.14 (2.16)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 142.62 (2.47) | 141.89 (2.12)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.23, ANCOVA
Statistical Analysis 2: Comparison: Cunermuspir; Test type: Other; p = 0.18, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; Blood sodium concentration between baseline and day 28 in the Placebo group; Test type: Other; p = 0.01, t-test, 2 sided

28. Secondary Outcome: Potassium
Description: changes in plasma potassium are reported in units of mmol per liter, reference value 3.5-5.4 mmol per liter, bloodbook.com
Time Frame: baseline and 28 days after enrollment
Population: The study sponsor is of the opinion that these participants were dehydrated when they started the study. They were instructed to drink more water. Three of the 56 that started the study were lost to followup or withdrew.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mmol/L
  baseline | 4.86 (0.45) | 4.84 (0.45)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 4.44 (0.43) | 4.39 (0.39)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.58, ANCOVA
Statistical Analysis 2: Comparison: Cunermuspir; comparison of blood potassium concentration upon enrollment and day 28 in the Cunermuspir participants; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; comparison of blood potassium concentrations from enrollment to day 28 in participants in the Placebo arm; Test type: Other; p < 0.001, t-test, 2 sided

29. Secondary Outcome: Chloride
Description: changes in plasma chloride are reported in uits of mmol per liter The reference range is 98-106 mmol per liter, bloodbook.com
Time Frame: baseline and 28 days after enrollment
Population: Enrollment pre-screening values are taken as the baseline. The study sponsor was of the opinion that these participants started the study dehydrated. Of the original 56 three were lost to followup or withdrew.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
mmol/L
  baseline | 106.14 (2.12) | 106.43 (2.27)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 105.08 (2.23) | 105.15 (1.99)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.87, ANCOVA
Statistical Analysis 2: Comparison: Cunermuspir; comparison between baseline and day 28 chloride concentrations in the Cunermuspir group; Test type: Other; p = 0.003, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; comparison of blood chloride concentrations between baseline and day 28 in Placebo Arm participants; Test type: Other; p = 0.003, t-test, 2 sided

30. Secondary Outcome: Bilirubin
Description: changes in total bilirubin are reported in units of micro moles per liter. Direct: up to 0.4 mg/dL, Total: up to 1.0 mg/dL bloodbook.com, Converts to 6.84-17.1 micro moles per liter. https://unitslab.com/node/37
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: micromol/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
micromol/L
  baseline | 11.0 (5.9) | 9.3 (3.5)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 11.2 (5.9) | 9.9 (4.3)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Bilirubin concentrations between Placebo and Cunermuspir compared at day 28; Test type: Other; p = 0.36, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cunermuspir; comparison of bilirubin concentrations between baseline and day 28 in the Cunermuspir Arm; Test type: Other; p = 0.72, Wilcoxon (Mann-Whitney); Wilcoxon Signed-Rank
Statistical Analysis 3: Comparison: Placebo; bilirubin concentrations compared between baseline and Day 28 in the Placebo Arm; Test type: Other; p = 0.35, Wilcoxon (Mann-Whitney)

31. Secondary Outcome: ALT
Description: changes in the liver enzyme alanine aminotransferase (ALT) in the blood are reported as units per liter Reference range 1 - 21 units/L bloodbook.com
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
U/L
  baseline | 27.6 (12.8) | 28.5 (16.3)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 28.2 (15.5) | 28.4 (15.4)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Test type: Other; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cunermuspir; comparison between baseline and day 28 values in Cunermuspir group; Test type: Other; p = 0.4, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo; comparison between baseline and day 28 values for the Placebo Arm; Test type: Other; p = 0.8, Wilcoxon (Mann-Whitney)

32. Secondary Outcome: AST
Description: changes in the liver enzyme aspartate aminotransferase (AST) in the blood are reported as units per liter Reference range 7 - 27 units/L bloodbook.com
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
U/L
  baseline | 23.0 (4.9) | 23.1 (6.3)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 24.2 (6.2) | 25.8 (9.5)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; comparison of AST enzyme activity in blood on day 28 between Cunermuspir and Placebo; Test type: Other; p = 0.62, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cunermuspir; baseline to day 28 comparison; Test type: Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo; baseline to day 28 comparison of AST activity in Placebo group; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney)

33. Secondary Outcome: GGT
Description: changes in the liver enzyme gamma-glutamyl transferase in the blood are reported as units per liter
Time Frame: baseline and 28 days after enrollment
Population: as for outcome 9
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
U/L
  baseline | 20.9 (13.6) | 28.6 (36.6)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 24.0 (18.1) | 25.6 (23.0)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; comparison between placebo and Cunermuspir at day 28; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney) — Comparison of GGT activities in blood of two arms: Cunermuspir and Placebo on Day 28
Statistical Analysis 2: Comparison: Cunermuspir; Comparison of GGT activities in participants' blood at baseline and on day 28; Test type: Other; p = 0.01, Wilcoxon Signed Rank
Statistical Analysis 3: Comparison: Placebo; Comparison of GGT activity in blood between Placebo Arm participants at baseline and on day 28; Test type: Other; p = 0.97, Wilcoxon Signed-Rank

34. Secondary Outcome: Copper
Description: changes in copper concentration in the blood are reported in units of micro moles per liter
Time Frame: baseline and 28 days after enrollment
Population: Of the 56 enrolled in the study three were lost to followup or dropped out.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cunermuspir | Placebo
Number analyzed (Participants) | 28 | 28
U/L
  baseline | 16.18 (2.42) | 17.62 (2.51)
  day 28: number analyzed (Participants) | 26 | 27
  day 28 | 16.6 (2.8) | 17.57 (2.89)
Statistical Analysis 1: Comparison: Cunermuspir vs Placebo; Between group comparisons were made using ANCOVA; Test type: Other; p = 0.03, ANCOVA
Statistical Analysis 2: Comparison: Cunermuspir; comparison of baseline with day 28; Test type: Other; p = 0.10, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo; comparison between baseline and day 28 serum copper concentrations in the Placebo Arm; Test type: Other; p = 0.89, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 28 days
Description: All treatment--emergent adverse events (AEs) are listed and MedDRA--coded to obtain the MedDRA Preferred Term and Organ System ("body system"). The nature, incidence, severity and causality were AEs were summarized in a frequency table, by body system and treatment. The proportion of subjects experiencing one or more AEs were compared between groups, separately for each body system and for all AEs combined.
Arm/Group | Cunermuspir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 6/26 | 7/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cunermuspir (N=26) | Placebo (N=27)
nasea (Gastrointestinal disorders) | 4 (4) | 3 (3) — also includes upset stomach, dry mouth, and dry mouth
seasonal respiratory infections (Infections and infestations) | 2 (2) | 4 (5) — includes sinusitis, common cold, and flu
moderate dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
head ache (Nervous system disorders) | 2 (2) | 1 (1) — the study investigators concluded that on of the two head ache in the Cunermuspir Arm may have been related to the study product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study PI (Dale Wilson) retired soon after the study was completed. KGK Synergize has undergone reorganization as KGK Science. The original intent was to publish the study results in a peer review journal.